CLINICAL TRIAL: NCT00098462
Title: A Phase I/II Trial of ZD1839 (Iressa®) and Rapamycin (Rapamune) in Patients With Advanced Non Small Cell Lung Cancer
Brief Title: Gefitinib and Sirolimus in Treating Patients With Recurrent or Refractory Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawn as study never opened
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000401501; UCLA-0407057-01; ZENECA-IRUSIRES0281
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Sirolimus

INTERVENTIONS:
Drug: gefitinib
Drug: sirolimus

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as sirolimus, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sometimes when chemotherapy is given, it does not stop the growth of tumor cells. The tumor is said to be resistant to chemotherapy. Giving gefitinib together with sirolimus may reduce drug resistance and allow the tumor cells to be killed.

PURPOSE: This phase I/II trial is studying the side effects and best dose of sirolimus when given with gefitinib and to see how well they work in treating patients with recurrent or refractory stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of sirolimus when combined with gefitinib in patients with recurrent or refractory stage IIIB or IV non-small cell lung cancer.

Secondary

* Determine the overall response rate (complete response [CR] and partial response [PR]) in patients treated with this regimen.
* Determine the disease control rate (CR, PR, and stable disease) in patients treated with this regimen.
* Determine the time to progression and overall survival of patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: This is an open-label, phase I, dose-escalation study of sirolimus followed by a phase II study.

* Phase I: Patients receive oral gefitinib once daily and oral sirolimus once daily on days 1-28. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of sirolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive gefitinib and sirolimus as in phase I at the MTD. Quality of life is assessed at baseline, day 1 of each course, and then at 1 month post-progression.

Patients are followed every 9 weeks. Patients withdrawn from study treatment without evidence of disease progression are followed every 6 weeks until disease progression.

PROJECTED ACCRUAL: A total of 25 patients (11 for phase I and 14 for phase II) will be accrued for this study within 8.3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer

  * Stage IIIB or IV disease
* Recurrent or refractory disease

  * Received ≥ 1 prior platinum-containing chemotherapy regimen
* Unidimensionally measurable disease that has not been irradiated
* No newly diagnosed untreated brain metastases or spinal cord compression
* Paraffin-embedded tumor tissue or slides available

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Adequate bone marrow function
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Adequate hepatic function
* No severe or uncontrolled hepatic disease

Renal

* Adequate renal function
* Creatinine ≤ 3.0 times upper limit of normal
* No severe or uncontrolled renal disease

Cardiovascular

* Adequate cardiac function
* No severe or uncontrolled cardiac disease
* No uncontrolled hyperlipidemia

Pulmonary

* No unstable or uncompensated respiratory disease
* No clinically active interstitial lung disease

  * Patients with chronic stable radiographic changes who are asymptomatic are eligible

Gastrointestinal

* Able to take oral medication
* No gastrointestinal condition (e.g., peptic ulcer disease) that would affect absorption

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious infection
* No known severe hypersensitivity to gefitinib or any of its excipients
* No other malignancy within the past 5 years except treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No other severe or uncontrolled systemic disease
* No significant clinical disorder or laboratory finding that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 14 days since prior biologic therapy
* No prior cetuximab, panitumumab, or bevacizumab

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior cytotoxic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* More than 3 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Recovered from prior oncologic or other major surgery
* No prior gastrointestinal surgery affecting absorption
* No concurrent surgery, including ophthalmic surgery, during and for 1 week after study treatment

Other

* Recovered from all prior therapy
* More than 30 days since prior investigational agents
* No other prior HER1/epidermal growth factor receptor axis agents, including the following:

  * Gefitinib
  * Erlotinib
  * CI-1033
  * Lapatinib
* No other prior vascular endothelial growth factor axis agents, including the following:

  * ZD6474
  * Vatalanib
* No concurrent CYP3A4 inducers, including the following:

  * Phenytoin
  * Carbamazepine
  * Rifampin
  * Phenobarbital
  * Barbiturates
  * Hypericum perforatum (St. John's wort)
* No other concurrent systemic treatment for the malignancy
* No concurrent bisphosphonates for symptomatic bone metastases
* No concurrent systemic retinoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-10

PRIMARY OUTCOMES:
Maximum tolerated dose (Phase I)

SECONDARY OUTCOMES:
Overall response (complete response [CR] and partial response [PR]) as measured by RECIST criteria
Disease control rate (CR, PR, and stable disease) correlated with smoking history
Time to tumor progression and overall survival
Quality of life as assessed by the Functional Assessment of Cancer Therapy-Lung (FACT-L)
Lung cancer subscale from FACT-L

CONTACTS AND LOCATIONS:
Overall Officials: Fairooz F. Kabbinavar, MD, Study Chair — Jonsson Comprehensive Cancer Center